Official Title PANOVA-3: Effect of Tumor Treating

of the study Fields (TTFields, 150 kHz) as Front-Line

**Treatment of Locally-advanced Pancreatic** 

**Adenocarcinoma Concomitant With** 

**Gemcitabine and Nab-paclitaxel** 

**NCT** number

**Document** 

**Date** 

NCT03377491

October 16, 2024

Study ID:

# **Statistical Analysis Plan**

# Novocure GmbH EF-27

PANOVA-3: Pivotal, randomized, open-label study of Tumor Treating Fields (TTFields, 150kHz) concomitant with gemcitabine and nab-paclitaxel for front-line treatment of locally-advanced pancreatic adenocarcinoma

Study ID:

Document Version:

Document Date:

Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

# Study ID:

# **Table of Contents**

| 1. | | Soul | rce Documents | 6 |
|----|-----|--------|-------------------------------------------------|----|
| 2. | | Prot | ocol Details | 6 |
| | 2.1 | St | udy Objectives | ε |
| | 2. | 1.1 | Primary Objectives | 6 |
| | 2. | 1.2 | Secondary Objectives | ε |
| | 2.2 | O۱ | verall Study Design | 7 |
| | 2.3 | Sa | ample Size and Power | 9 |
| 1. | | Effic | acy and Safety Variables | 9 |
| | 3.1 | Pr | imary Efficacy Endpoint | 9 |
| | 3.2 | Se | econdary Efficacy Endpoints | 10 |
| | 3.3 | Sa | nfety Variables | 13 |
| 4 | P | harm | acokinetic/Pharmacodynamic variables | 15 |
| 5 | Α | nalys | sis populations | 16 |
| | 5.1 | In | tent-to-treat Population | 16 |
| | 5.2 | М | odified Intent-to-treat Population | 16 |
| | 5.3 | Sa | afety Population | 16 |
| 6 | D | ATA | Handling | 16 |
| | 6.1 | Tii | me points and Visit Windows | 16 |
| | 6.2 | На | andling of Dropouts, Missing Data, and Outliers | 17 |
| 7 | S | tatist | tical Methods | 17 |
| | 7.1 | Ge | eneral Principles | 17 |
| | 7.2 | Su | ubject Disposition and Data Sets Analyzed | 19 |
| | 7.3 | Pr | otocol Deviations | 20 |
| | 7.4 | De | emographics and Other Baseline Characteristics | 20 |
| | 7. | 4.1 | Medical History | 21 |
| | 7. | 4.2 | Previous and Concomitant Medications | 21 |
| | 7.5 | Ef | ficacy | 22 |
| | 7. | 5.1 | Primary Efficacy Analysis | 22 |
| | 7. | 5.2 | Secondary Efficacy Analysis | 23 |
| | 7. | 5.3 | Sensitivity Analysis | 27 |

Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

| CL J. | . ID. |
|-------|-------|
| Stud | v iD: |

| Subgroup Analysis | 27 |
|------------------------------------------|-------------------|
| Safety | 28 |
| Extent of Exposure and device compliance | 28 |
| Adverse Events | 30 |
| Laboratory Evaluations | 31 |
| Vital Signs | 32 |
| • | |
| | Subgroup Analysis |

Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

| Stu | dv | ID | 1 |
|-------|----|----|---|
| ) Stu | uv | 1L | , |

# **Reviewers**

The following reviews of the SAP were conducted:

| Name and Title | Role | Version Last | Company/ |
|----------------|------|--------------|--------------|
| | | Reviewed | Organization |

Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Study ID:

# **Glossary of Abbreviations**

| Abbreviation | Term |
|--------------|------------------------------------------------------------|
| AE | Adverse Event |
| ADE | Adverse Device Effect |
| CA | Competent Authority |
| CA 19-9 | Carbohydrate Antigen 19-9 |
| CI | Confidence Interval |
| Cm | Centimeter |
| CR | Complete Response |
| CRF | Case Report Form |
| СТ | Computed Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DMC | Data and Monitoring Committee |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| EORTC | European Organization for Research and Treatment of Cancer |
| FDA | Food and Drug Administration |
| ITT | Intent to Treat |
| mITT | Modified Intent to Treat |
| LDH | Lactatdehydrogenase |
| MRI | Magnetic Resonance Imaging |
| NCI | National Cancer Institute |
| ORR | Objective Response Rate |
| OS | Overall Survival |
| PFS | Progression Free Survival |
| PR | Partial Response |
| PT | Preferred Term |
| QLQ C-30 | EORTC's Quality of life Questionnaire C-30 |
| QLQ PAN26 | Quality of life questionnaire Pancreatic Cancer Module |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SAF | Safety Population |
| SOC | Standard of Care |
| TEAEs | Treatment-emergence adverse events |
| TTFields | Tumor Treating Fields |
| VAS | Visual Analogue Scale |


Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Study ID:

#### 1. SOURCE DOCUMENTS

The Statistical Analysis Plan (SAP) was written based on the following documentation:

| Document | Date | Version |
|----------|------|---------|
| Protocol | | |
| eCRF | | |

#### 2. PROTOCOL DETAILS

# 2.1. Study Objectives

# 2.1.1. Primary Objectives

To determine if TTFields concomitant with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients prolongs the overall survival of patients, compared to chemotherapy treatment alone.

# 2.1.2. Secondary Objectives

- To determine if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients prolongs the progression-free survival of patients, compared to chemotherapy treatment alone.
- To determine if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients prolongs the local progression-free survival of patients, compared to chemotherapy treatment alone.
- 3. To determine if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients leads to a higher rate of objective response rate, compared to chemotherapy treatment alone.
- 4. To determine if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients leads to a higher 1-year survival rate, compared to chemotherapy treatment alone.
- 5. To assess if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients affects the quality of life of patients, compared to chemotherapy treatment alone.
- 6. To evaluate if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients


Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Study ID:

prolongs the pain-free survival of patients, compared to chemotherapy treatment alone.

- 7. To determine if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients prolongs the puncture-free survival of patients, compared to chemotherapy treatment alone.
- 8. To determine if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients increases the probability of the cancer becoming resectable (with a curative intention), compared to chemotherapy treatment alone.
- 9. To determine if TTFields in combination with gemcitabine and nab-paclitaxel in the first line treatment of unresectable, locally advanced pancreatic cancer patients is a safe treatment compared to chemotherapy treatment alone.

#### 2.2. Overall Study Design

This is a pivotal, randomized, open-label, two-arm, multicenter study. This randomized study is designed to test the efficacy and safety of gemcitabine and nab-paclitaxel, with or without TTFields, using the NovoTTF-200T System as a front-line therapy for locally-advanced pancreatic adenocarcinoma patients. The study population are the patients with unresectable, locally-advanced adenocarcinoma of the pancreas, and with ECOG 0-2. Patients will be stratified as below:



- 1. Arm I: Patients receive TTFields using the NovoTTF-200T System together with gemcitabine and nab-paclitaxel.
- 2. Arm II: Patients receive gemcitabine and nab-paclitaxel alone.

| | COMPTENDENT | D 7 C 27 |
|----------------|--------------|-----------------------------------------|
| | | 1 2 3 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 |
| Document Date: | | |

| Sponsor Name. Novocure Ltd. | 0: 1 10 |
|-----------------------------|-----------|
| Sponsor Protocol ID: EF-27 | Study ID: |

Patients on both arms should also receive the best supportive care available at each site. Following progression patients may be offered standard pancreatic cancerdirected therapy and salvage therapy based on local practice at each site. Treatment may continue post-radiation therapy if radiation therapy is applied prior to local disease progression, as long as the skin has recovered from the radiation therapy according to the study investigator. Treatment may continue post-surgical resection if patient becomes resectable, as long as the skin has recovered from the surgical wounds according to the study investigator.

The overall schedule of the study is as follows:




Document Date:

| Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27 | Study ID: |
|---|---|
| - Sportson (1910-00) 25 Et 27 | otaay 15. |
| 2.3. Sample Size and Power | |
| 3. EFFICACY AND SAFETY VARIABLES | |
| 3.1. Primary Efficacy Endpoint | |
| Overall survival (OS) of patients treated with TTFields con<br>and nab-paclitaxel in the first line treatment of unre<br>pancreatic cancer patients, compared to overall survival<br>chemotherapy alone. | sectable, locally advanced |
| OS will be measured from the date of randomization to the | e date of death (in months). |


Document Date:

| Statistical Analysis Plan Sponsor Name: NovoCure Ltd. |
|---|
| Sponsor Protocol ID: EF-27 Study ID: |
| 3.2. Secondary Efficacy Endpoints |
| 3.2.1. Progression-free survival (PFS) |
| PFS of patients treated with TTFields concomitant with gemcitabine and nab-paclitaxel, compared to that of patients treated with chemotherapy alone, using the RECIST V1.1 Criteria. |
| Progression-free survival is defined as the time from the date of randomization until the date of disease progression for the entire body according to RECIST Criteria Version 1.1 or death (by any cause in the absence of progression). |
| 3.2.2. Local progression-free survival |
| Local disease progression is defined as Progressive Disease per revised RECIST |
| version 1.1 in the absence of distant metastasis |
| Local progression-free survival is defined as the time from the date of |

randomization until the date of local disease progression as defined above (by any

 Document Date:

| Sponsor Name: NovoCure Ltd.<br>Sponsor Protocol ID: EF-27 | Study ID: |
|---|---|
| cause in the absence of local disease progression) | or death |
| 3.2.3. Objective response rate (ORR) | |
| The objective response to the tumor will be assess to the revised RECIST Criteria V1.1. Objective responserion of patients with best response of partial response (CR) between the time of randomization progression or death. | ponse rate is defined as the<br>Il-response (PR) or complete |
| progression of death. | |
| 3.2.4. One-year survival rate | |
| One-year survival rate of patients treated with TTI gemcitabine and nab-paclitaxel in the first line treadvanced pancreatic cancer patients, compared to patients treated with chemotherapy alone. | atment of unresectable, locally |
| 3.2.5. Quality of life | |
| Quality of life of patients are assessed using the E the PAN26 addendum. | ORTC QLQ C30 questionnaire with |


Document Date:

| Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27 | Study ID: |
|---|---|
| Sponsor Frotocor IB. El 27 | Study ID. |
| 2.2.6. Dain for a security I | |
| 3.2.6. Pain-free survival | |
| Pain-free survival measures the duration between the greater than or equal to points increase, which baseline measurement of a patient self-reported visual recorded or death, whichever occurs first. | means pain increase, from |
| | _ |
| _ | |

# 3.2.7. Puncture-free survival

Puncture-free survival will be measured as the duration between randomization until the first need for paracentesis as data collected on the ascitic fluid drainage


Document Date:

Sponsor Name: NovoCure Ltd. Study ID: Sponsor Protocol ID: EF-27 eCRF or death, whichever occurs first. 3.2.8. Resectability rate Resectability rate will be measured as the percentage of patients whose tumors were deemed resectable. PT terms MEDDRA codes 3.3. Safety Variables 3.3.1. Extend of Exposure 3.3.1.1. Extend exposure to NovoTTF-200T Extend of exposure to NovoTTF-200T will be summarized descriptively for the patients who randomized to the NovoTTF-200T arm as:


Document Date:

| Sponsor N | Statistical Analysis Plan<br>Name: NovoCure Ltd. |
|---|---|
| | Protocol ID: EF-27 Study ID: |
| 3.3.1.2 | . Exposure to Standard of Care |
| | d of care in this study contains two drugs: Nab-paclitaxel and Gemcitabine a drug, the following variables will be determined: |
| 3.3.2. <i>A</i> | Adverse Events (AEs) |
| dictiona<br>immedia | erse events (AEs) recorded on the eCRF will be coded using the MedDRA ry [Version 20.1-23.0]. The adverse event reporting period will begin ately following randomization. Adverse events will be collected until last study p visit and for following treatment termination |
| the first | ent-emergence adverse events (TEAEs) are events with start date on or after<br>date of any study treatment (including SOC or TTFields), or events with star<br>or to the date of first treatment whose severity worsens on or after the date<br>atment. |
| | nent of AE severity will be based on the National Cancer Institute (NCI necession) near the Terminology Criteria for Adverse Events (CTCAE) version 4.03. |
| possible | ationship between an AE and study device is assessed as definite, probable, unlikely, or none. A device-related AE is an AE considered by the ator as definitely, possibly, or probably related to study device. |
| 3.3.3. L | aboratory Evaluations |

Document Date:

 Sponsor Name: NovoCure Ltd.

Study ID: Sponsor Protocol ID: EF-27



# 3.3.4. Vital Signs

The following vital signs will be evaluated

# 3.3.5. Physical Examination

Physical examination assessments including will be performed according to the study schedule.

# 4. PHARMACOKINETIC/PHARMACODYNAMIC VARIABLES

Not applicable.

 Document Date:

Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Study ID:


#### 5. ANALYSIS POPULATIONS

#### 5.1. Intent-to-treat Population

The Intent-to-treat (ITT) will consist of all randomized subjects regardless of treatment receipt. ITT subjects are analyzed according to their randomized treatment.

# 5.2. Modified Intent-to-treat Population

The Modified Intent-to-treat (mITT) will consist of all patients who received at least one complete cycle of study treatments.

#### 5.3. Safety Population

The safety population (SAF) will include all patients who received any amount of study Standard of Care drugs or TTFields in the experimental arm, and any amount of study Standard of Care drugs in the control arm.

#### 6. DATA HANDLING

Document Date:

#### 6.1. Time points and Visit Windows

| · | |
|---------------------------------------|----|
| | I, |


Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Study ID:

# 6.2. Handling of Dropouts, Missing Data, and Outliers



# 7. STATISTICAL METHODS

# 7.1. General Principles

| All data | processing, | summarization | and | analyses will | be performed using | |
|---|---|---|---|---|---|---|
| | | | | of the $SAS^{\scriptscriptstyle{(\! g)}}$ | statistical software p | oackage. |


Document Date:

Sponsor Name: NovoCure Ltd.



**Table 1** Statistical Analysis General Principles

| Principle | Value |
|-----------|-------|


Document Date:

Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Document Date:

| cu. | |
|-----|-----------|
| | Study ID: |

| Principle | Value |
|-----------|-------|

# 7.2. Subject Disposition and Data Sets Analyzed




Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Study ID:



#### 7.3. Protocol Deviations



# 7.4. Demographics and Other Baseline Characteristics

Demographic and baseline characteristics will be listed and summarized by treatment group and overall for ITT populations.

Standard descriptive statistics will be presented for the continuous variable of:



The total counts and percentages of subjects will be presented for the categorical variables of:

- Gender (Female, Male);
  - Childbearing potential (Yes, No), if female;
  - If no, reason (Surgically sterile, Post-menopausal, Other).


Document Date:

| Statistical Analysis Plan | |
|----------------------------------------------------------|-----------|
| Sponsor Name: NovoCure Ltd. | |
| Sponsor Protocol ID: EF-27 | Study ID: |
| • Race | |
| <ul> <li>Ethnicity</li> </ul> | |
| Cincolla socialization | |
| <ul> <li>Cigarette smoking status</li> </ul> | |
| <ul> <li>ECOG performance status</li> </ul> | |
| Region | |
| 7.4.1. Medical History | |
| Madical bistory will be reded using the Madical Distings | |

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) [Version 20.1-23.0]. All medical history will be listed, and the number and percentage of subjects with any medical history will be summarized for safety population by system organ class (SOC) and preferred term (PT) for each treatment group and overall.

#### 7.4.2. Previous and Concomitant Medications

A listing of prior treatments and procedures for pancreatic cancer will be presented.

Medications received prior to or concomitantly with treatment will be coded using the WHO Drug Dictionary [March 2016], Anatomical Therapeutic Chemical (ATC) Classification codes.

Prior medications and concomitant medications are defined as follows:

 Document Date:

| Statistical Analysis Plan |
|---|
| Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27 Study ID: |
| 7 E Efficacy |
| 7.5. Efficacy |
| 7.5.1. Primary Efficacy Analysis |
| The primary endpoint is to compare overall survival (OS) of patients treated with TTFields concomitant with standard of care of chemotherapy (SOC) versus patient treated with SOC alone. |
| The null hypothesis is that the OS is the same in the two study groups, i.e., hazar ratio=1. The alternative hypothesis is that the OS is not the same, i.e., hazar ratio $\pm 1$ . |
| The primary endpoint will be summarized using Kaplan-Meier (KM) estimate. The treatment difference will be tested using a in ITT population in order to allow for two efficacy analyses of the primary endpoint (interim analysis and final analysis |


Document Date:

| Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27 | Study ID: |
|---|---|
| 7.5.2. Secondary Efficacy Analysis | |
| The secondary endpoint of progression free survival primary endpoint of OS met its significance level. Thus, the enbe allocated to the progression free survival endpoint and no a made for multiple hypothesis testing. | tire alpha of 0.05 will |
| 7.5.2.1. Progression-free Survival | |
| test at an alpha level of 0.05 wi<br>the difference of progression-free survival between the patients<br>concomitant with SOC and the patients treated with SOC alo | treated with TTFields |
| The median, 25th and 75th percentiles of progression-free survible estimated using the Kaplan-Meier method for the two tr | |


Document Date:

| Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27 Study ID: |
|---|
| 7.5.2.2. Local Progression-free Survival |
| test at an alpha level of 0.05 will be used to evaluate if the local PFS will be significantly greater in the TTFields + SOC arm than in the SOC alone arm |
| The median, 25th and 75th percentiles of local progression-free survival with 95% CIs will be estimated using the Kaplan-Meier method for the two treatment groups |
| 7.5.2.3. One Year Overall Survival Rate |
| One-year overall survival (OS) rate is the proportions of patients who are alive at 12 months in each arm of the study. The Kaplan-Meier estimates of survival at Year 1 will be presented with number at risk, number with events, and estimated survival probability. |
| The one-year OS rates will be compared using |
| 7.5.2.4. Objective Radiological Response Rate |
| Objective radiological response rate (ORR) and its two-sided 95% confidence interval which is based on presented. |


Document Date:

Statistical Analysis Plan Sponsor Name: NovoCure Ltd. Study ID: Sponsor Protocol ID: EF-27 **7.5.2.5. Quality of Life Questionnaire Scores** Scores from 0-100 will be derived for all multi-item or single item scales of the EORTC QLQ-C30 and QLQ-PAN26.


Document Date:

Table 2. Clinically meaningful change and categories



#### 7.5.2.6. Pain-free Survival



#### 7.5.2.7. Puncture-free Survival

A test at an alpha level of 0.05 will be used to evaluate if TTFields + SOC prolongs the puncture-free survival of patients, compared to SOC


Document Date:

Sponsor Name: NovoCure Ltd. Study ID: Sponsor Protocol ID: EF-27 treatment alone The median, 25th and 75th percentiles of puncture-free survival with 95% CIs will be estimated using the Kaplan-Meier method for the two treatment groups 7.5.2.8. Resectability Rate , which is based on the Resectability rate and its will be presented. The resectability rate between the patients treated with TTFields concomitant with SOC and the patients treated with SOC alone will be compared using assuming the TTFields plus the chemotherapy arm would have a higher resectability rate than the chemotherapies alone arm. 7.5.3. Sensitivity Analysis 7.5.4. Subgroup Analysis


Document Date:

**Statistical Analysis Plan** Sponsor Name: NovoCure Ltd. Study ID: Sponsor Protocol ID: EF-27 7.6. Safety

# 7.6.1. Extent of Exposure

# 7.6.1.1. Exposure to NovoTTF-200T

usage will be summarized descriptively for the patients who randomized to the NovoTTF arm. The total counts and percentages of subjects will be presented for the categorical variables of:

 Document Date:

Sponsor Name: NovoCure Ltd.
Sponsor Protocol ID: EF-27

Study ID:

# 7.6.1.2. Exposure to Standard of Care

Standard of care in this study contains two drugs: Nab-paclitaxel and Gemcitabine. For each drug, total dose administered, and duration of exposure will be summarized by each treatment group in safety population using continuous descriptive statistics. Duration of exposure will be calculated as the total number of weeks from the first date of dose to the last date of dose plus 1 day:




Document Date:

Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Document Date:

Study ID:


# 7.6.2. Adverse Events

An overview table will summarize the number and percentage of subjects with at least one of the following AEs by treatment group and overall, where subjects with more than one AE in a particular category are counted only once in that category:

| A similar overall table summarizing treatment emergent AE will also be created. |
|---|
| The number and percentage of subjects reporting each AE will be summarized |
| for the Safety population. Tables |
| will be sorted alphabetically by SOC. PTs will be sorted by descending overall total |
| The following summaries will be produced: |


Sponsor Name: NovoCure Ltd. Study ID: Sponsor Protocol ID: EF-27 7.6.3. Laboratory Evaluations Data for the following analyses recorded in the eCRF will be listed and summarized

 Document Date:

Statistical Analysis Plan Sponsor Name: NovoCure Ltd. Study ID: Sponsor Protocol ID: EF-27 All laboratory data will be reported in International System of Units (SI) units. Laboratory data will be summarized for the Safety population. For each laboratory analytic, 7.6.4. Vital Signs The following vital signs Vital signs data and changes from baseline in vital signs will be summarized for the Safety population. 7.6.5. Physical Examination Physical examination data will be listed.


Document Date:

Sponsor Name: NovoCure Ltd.
Sponsor Protocol ID: EF-27
Study ID:

# 7.7. Interim Analysis

| One interim analysis will be performed on the OS data available |
|-----------------------------------------------------------------|

#### 8. CHANGES IN PLANNED ANALYSIS

#### 9. REFERENCES

- 1. Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer. 45:228-247. doi:10.1016/j.ejca.2008.10.026.
- 2. Hammel P, Huguet F, van Laethem J-L, et al. Effect of Chemoradiotherapy vs Chemotherapy on Survival in Patients With Locally Advanced Pancreatic Cancer Controlled After 4 Months of Gemcitabine With or Without Erlotinib. JAMA. 2016;315(17). doi:10.1001/jama.2016.4324.
- 3. Von Hoff DD, Ervin T, Arena FP, et al. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013;369(18):1691-1703. doi:10.1056/NEJMoa1304369.
- 4. Anne AE, Paul K, Mithat G, et al. Psychometric Validation of the EORTC QLQ-PAN26 Pancreatic Cancer Module for Assessing Health Related Quality of Life after Pancreatic Resection. J Pancreas. 2017; 1027;18(1):19-25


Document Date:

Sponsor Name: NovoCure Ltd. Sponsor Protocol ID: EF-27

Study ID:

# 10. APPENDICES

# 10.1. Scoring algorithm for the EORTC-QLQC30



Sponsor Name: NovoCure Ltd. Study ID: Sponsor Protocol ID: EF-27


Document Date:

Sponsor Name: NovoCure Ltd.

Study ID: Sponsor Protocol ID: EF-27



# 10.2. Scoring algorithm for the PAN26



**CONFIDENTIAL**  Document Date:

Sponsor Name: NovoCure Ltd.
Sponsor Protocol ID: EF-27

Study ID:


Document Date: